CLINICAL TRIAL: NCT06330246
Title: Oxalobacter Formigenes Colonization in Calcium Oxalate Kidney Stone Formers
Brief Title: O. Formigenes Colonization in Calcium Oxalate Kidney Stone Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sonia Fargue, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300005280-OCK; R01DK137784 (NIH)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stone; Kidney Calculi; Urolithiasis; Urolithiasis, Calcium Oxalate; Nephrolithiasis; Nephrolithiasis, Calcium Oxalate; Oxalate Urolithiasis; Oxaluria
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis, Calcium Oxalate; Nephrolithiasis; Hyperoxaluria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- colonization with Oxalobacter formigenes (Experimental): Colonization with a live preparation of Oxalobacter formigenes, strain OxCC13.
  Interventions: Dietary Supplement: Low oxalate fixed diets pre-colonization; Dietary Supplement: Moderately high oxalate fixed diets pre-colonization; Dietary Supplement: Colonization with Oxalobacter formigenes; Dietary Supplement: Low oxalate fixed diets post-colonization; Dietary Supplement: Moderately high oxalate fixed diets post-colonization

INTERVENTIONS:
Dietary Supplement: Low oxalate fixed diets pre-colonization — 4 days of fixed eucaloric diet with low oxalate (< 60 mg/day), normal calcium (600-1000 mg/day)
Dietary Supplement: Moderately high oxalate fixed diets pre-colonization — 4 days of fixed eucaloric diet with moderately high oxalate (250-300 mg/day), normal calcium (600-1000 mg/day)
Dietary Supplement: Colonization with Oxalobacter formigenes — Ingestion of live Oxalobacter formigenes
Dietary Supplement: Low oxalate fixed diets post-colonization — 4 days of fixed eucaloric diet with low oxalate (< 60 mg/day), normal calcium (600-1000 mg/day)
Dietary Supplement: Moderately high oxalate fixed diets post-colonization — 4 days of fixed eucaloric diet with moderately high oxalate (250-300 mg/day), normal calcium (600-1000 mg/day)

SUMMARY:
The goal of this trial is to test if colonization with the gut bacteria Oxalobacter formigenes leads to a reduction in urinary oxalate excretion in patients with calcium oxalate kidney stone disease.

The study will recruit adult participants with a history of calcium oxalate kidney stones who are not colonized with Oxalobacter formigenes.

Participants will

* ingest fixed diets containing low and moderately high amounts of oxalate for 4 days at a time
* collect urine, blood and stool samples during the fixed diets
* ingest a preparation of live Oxalobacter formigenes to induce colonization with Oxalobacter formigenes

DETAILED DESCRIPTION:
In this study the investigators propose to measure the excretion of urinary oxalate on a fixed diet with controlled amounts of oxalate, before and after inducing colonization with the gut bacteria Oxalobacter formigenes in individuals with a history of calcium oxalate kidney stones not already colonized with Oxalobacter formigenes.

Screening and Pre-colonization phase. Between the University of Alabama at Birmingham (UAB) and the University of Texas Southwestern Medical Center (UTSW), the study will enroll 40 individuals with a history of idiopathic calcium oxalate kidney (20 males/20 females). Screening will include stool colonization testing, blood complete metabolic profile, 24-hr urine specimens collected at home on self-selected diets and anthropometric measurements.

Participants will ingest a low-oxalate (<60 mg/day) fixed diet for 4 consecutive days and collect two 24-hr urines and a stool sample after 2 days of dietary equilibration, as well as one fasted blood sample on the last morning.

After a wash-out period of at least 1 week, participants will ingest a moderately high-oxalate (250-300 mg/day) fixed diet for 4 consecutive days and collect two 24-hr urines and a stool sample after 2 days of dietary equilibration, as well as one fasted blood sample on the last morning.

Colonization and Post-colonization phase. Participants will be colonized with Oxalobacter formigenes by ingesting a freshly thawed paste of live bacterial preparation of O. formigenes. They will collect a stool sample 1 week later to assess if colonization occured.

After confirmation of successful colonization, participants will ingest a low-oxalate (<60 mg/day) fixed diet for 4 consecutive days and collect two 24-hr urines and a stool sample after 2 days of dietary equilibration, as well as one fasted blood sample on the last morning.

After a wash-out period of at least 1 week, participants will ingest a moderately high-oxalate (250-300 mg/day) fixed diet for 4 consecutive days and collect two 24-hr urines and a stool sample after 2 days of dietary equilibration, as well as one fasted blood sample on the last morning.

Follow-up phase Participants will be followed up every 6 months to assess sustainability of colonization, provide a stool sample and answer a simple questionnaire. A 24-hr urine collection will be requested once a year after colonization, on the same moderately high oxalate diet diet after 2 days of dietary equilibration.

ELIGIBILITY:
Inclusion Criteria

* age 19-70 yrs
* Body Mass Index > 18.5 kg/m2
* First time or recurrent Calcium Oxalate stone former. Composition of most recent stone ≥ 50% calcium oxalate if available
* Not colonized with Oxalobacter formigenes
* Normal fasting serum electrolytes on comprehensive metabolic profile
* Willing to ingest fixed diets
* Willing to stop supplements (vitamins including vitamin C, calcium (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, probiotics) for 2 weeks before start and during fixed diet phases.
* If on medications for stone prevention (e.g. thiazides, citrate, allopurinol), stable dose regimen for at least 2 weeks prior to and during study

Exclusion Criteria

* Chronic Kidney Disease stage 4-5
* Primary hyperoxaluria
* Liver, endocrine or renal diseases (other than idiopathic Calcium Oxalate kidney stones) or any other condition that may influence the absorption, transport or urinary excretion of ions, which will compromise the interpretation of results, including: Cystic fibrosis, Cystinuria, Uric acid stone former, Nephrotic syndrome, Sarcoidosis, Renal tubular acidosis, Primary hyperparathyroidism, Neurogenic bladder, Urinary diversion
* Pregnancy or breast-feeding
* Incompatible dietary requirements with the study, food allergies or intolerance to any of the foods in study menus
* Active malignancy or treatment for malignancy within 12 months prior to screening
* Utilization of immunosuppressive medication
* Uncontrolled Hypertension or diabetes
* Diabetes type 1
* Current Colonization with Oxalobacter formigenes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in urinary oxalate excretion following colonization with Oxalobacter formigenes | 2 months
  Difference between urinary oxalate excretion on the moderately high oxalate diet pre-colonization and urinary oxalate excretion on the moderately high oxalate diet post-colonization

SECONDARY OUTCOMES:
Sustainability of colonization with Oxalobacter formigenes | 4 years
  duration of colonization after successful induction of colonization sith Oxalobacter formigenes

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Fargue, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UTSW, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No